CLINICAL TRIAL: NCT01455298
Title: Research of Infra Clinical Liver Injuries in Adult Patients Presented With Alpha-1 AT Deficiency
Brief Title: Liver Disease in Adults With Alpha-1 AT Deficiency
Acronym: LIDIA-A1AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2011.664
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2012-10

CONDITIONS: Alpha-1 AT Deficiency
Keywords: Alpha-1 AT deficiency; liver injury; Transient Elastography; FibroTest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transient elastography and fibrotest (Other)
  Interventions: Other: Transient Elastography and fibrotest

INTERVENTIONS:
Other: Transient Elastography and fibrotest — a Transient Elastography and an ultrasound are performed.

SUMMARY:
This cohort study will evaluate the prevalence of the infra clinical liver injuries among a group of adult patients presenting with Alpha-1 AT deficiency followed up in a large university hospital in Lyon, France.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Presenting an Alpha-1 AT deficiency (Alpha-1 AT level <0.8g/l at the time of diagnosis)

Exclusion Criteria:

* Patients presenting a liver disease not related to the Alpha-1 AT deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The prevalence of infra clinical liver injuries | At least one day depending on the schedule of the exams
  The prevalence of infra clinical liver injuries (lesions or liver abnormalities) in a cohort of adult patients presenting an Alpha-1 AT deficiency. Suspicion of fibrosis was defined as liver stiffness > 7.2kPa measured by transient elastography (TE).

SECONDARY OUTCOMES:
morphological liver complications description | At least one day depending on the schedule of the exams
  To describe all the morphological liver complications present at the moment of the investigation.
measure of biological parameters | At least one day depending on the schedule of the exams
  - To measure the biological parameters (as AST, ALT, GGT, total bilirubin, lymphocytes, platelets, FibroTest score) and radiological aspects (TE score, liver aspect evaluated by ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François MORNEX, PhD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant - Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Result] Guillaud O, Dumortier J, Traclet J, Restier L, Joly P, Chapuis-Cellier C, Lachaux A, Mornex JF. Assessment of liver fibrosis by transient elastography (Fibroscan(R)) in patients with A1AT deficiency. Clin Res Hepatol Gastroenterol. 2019 Feb;43(1):77-81. doi: 10.1016/j.clinre.2018.08.016. Epub 2019 Jan 3. PMID 30612958